CLINICAL TRIAL: NCT05826899
Title: A Stable Isotope Study in Young Iron-depleted Thai Women to Evaluate the Bioavailability of an Oat Protein-based Iron Delivery System
Brief Title: A Stable Isotope Study to Evaluate the Bioavailability of an Oat Protein-based Iron Delivery System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Rainforest Company (Industry)
Collaborators: Mahidol University (Other); Swiss Federal Institute of Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: RainforestCo
Record Dates: First submitted 2023-04-09; First posted 2023-04-24 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2023-11

CONDITIONS: Bioavailability
Keywords: oat protein; iron-depleted woman; stable isotope
MeSH Terms: interventions — Honey

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- oat protein-based iron delivery system1 (Active Comparator): Each subject will complete the six iron absorption studies in which they will receive supplemental iron doses of 4 mg iron from the six products: (i) Fe-oat 1 alone, (ii) Fe-oat 1 with 30 mL acai puree with honey, (iii) Fe-oat 2 alone, (iv) Fe-oat 2 with 30 mL acai puree with honey, (v) FeSO4 alone, (vi) FeSO4 with 30 mL acai puree and honey.
  Interventions: Other: 54Fe SO4; Other: 57Fe Oat-1; Other: 58Fe Oat-2; Other: 54 FeSO4 + Acai puree with honey; Other: 57Fe Oat-1 + Acai puree with honey; Other: 58Fe Oat-2 + Acai puree with honey
- oat protein-based iron delivery system2 (Active Comparator): Each subject will complete the six iron absorption studies in which they will receive supplemental iron doses of 4 mg iron from the six products: (i) Fe-oat 1 alone, (ii) Fe-oat 1 with 30 mL acai puree with honey, (iii) Fe-oat 2 alone, (iv) Fe-oat 2 with 30 mL acai puree with honey, (v) FeSO4 alone, (vi) FeSO4 with 30 mL acai puree and honey.
  Interventions: Other: 54Fe SO4; Other: 57Fe Oat-1; Other: 58Fe Oat-2; Other: 54 FeSO4 + Acai puree with honey; Other: 57Fe Oat-1 + Acai puree with honey; Other: 58Fe Oat-2 + Acai puree with honey
- oat protein-based iron delivery system3 (Active Comparator): Each subject will complete the six iron absorption studies in which they will receive supplemental iron doses of 4 mg iron from the six products: (i) Fe-oat 1 alone, (ii) Fe-oat 1 with 30 mL acai puree with honey, (iii) Fe-oat 2 alone, (iv) Fe-oat 2 with 30 mL acai puree with honey, (v) FeSO4 alone, (vi) FeSO4 with 30 mL acai puree and honey.
  Interventions: Other: 54Fe SO4; Other: 57Fe Oat-1; Other: 58Fe Oat-2; Other: 54 FeSO4 + Acai puree with honey; Other: 57Fe Oat-1 + Acai puree with honey; Other: 58Fe Oat-2 + Acai puree with honey
- oat protein-based iron delivery system4 (Active Comparator): Each subject will complete the six iron absorption studies in which they will receive supplemental iron doses of 4 mg iron from the six products: (i) Fe-oat 1 alone, (ii) Fe-oat 1 with 30 mL acai puree with honey, (iii) Fe-oat 2 alone, (iv) Fe-oat 2 with 30 mL acai puree with honey, (v) FeSO4 alone, (vi) FeSO4 with 30 mL acai puree and honey.
  Interventions: Other: 54Fe SO4; Other: 57Fe Oat-1; Other: 58Fe Oat-2; Other: 54 FeSO4 + Acai puree with honey; Other: 57Fe Oat-1 + Acai puree with honey; Other: 58Fe Oat-2 + Acai puree with honey
- oat protein-based iron delivery system5 (Active Comparator): Each subject will complete the six iron absorption studies in which they will receive supplemental iron doses of 4 mg iron from the six products: (i) Fe-oat 1 alone, (ii) Fe-oat 1 with 30 mL acai puree with honey, (iii) Fe-oat 2 alone, (iv) Fe-oat 2 with 30 mL acai puree with honey, (v) FeSO4 alone, (vi) FeSO4 with 30 mL acai puree and honey.
  Interventions: Other: 54Fe SO4; Other: 57Fe Oat-1; Other: 58Fe Oat-2; Other: 54 FeSO4 + Acai puree with honey; Other: 57Fe Oat-1 + Acai puree with honey; Other: 58Fe Oat-2 + Acai puree with honey
- oat protein-based iron delivery system6 (Active Comparator): Each subject will complete the six iron absorption studies in which they will receive supplemental iron doses of 4 mg iron from the six products: (i) Fe-oat 1 alone, (ii) Fe-oat 1 with 30 mL acai puree with honey, (iii) Fe-oat 2 alone, (iv) Fe-oat 2 with 30 mL acai puree with honey, (v) FeSO4 alone, (vi) FeSO4 with 30 mL acai puree and honey.
  Interventions: Other: 54Fe SO4; Other: 57Fe Oat-1; Other: 58Fe Oat-2; Other: 54 FeSO4 + Acai puree with honey; Other: 57Fe Oat-1 + Acai puree with honey; Other: 58Fe Oat-2 + Acai puree with honey

INTERVENTIONS:
Other: 54Fe SO4 — 4 mg of iron as FeSO4 labelled with 4 mg of 54Fe
Other: 57Fe Oat-1 — 4 mg of iron as 0.46 g Fe-oat 1 (Oat fibrils, ascorbic acid reduced) labelled with 57Fe
Other: 58Fe Oat-2 — 4 mg of iron as 0.46 g Fe-Oat 2 (Fe-Oat with NaOH) labelled with 58Fe.
Other: 54 FeSO4 + Acai puree with honey — 4 mg of iron as FeSO4 labelled with 4 mg of 54Fe given with 30 mL acai puree with honey.
Other: 57Fe Oat-1 + Acai puree with honey — 4 mg of iron as 0.46 g Fe-oat 1 (Oat fibrils, ascorbic acid reduced) labelled with 57Fe given with 30 mL acai puree with honey.
Other: 58Fe Oat-2 + Acai puree with honey — 4 mg of iron as 0.46 g Fe-Oat 2 (Fe-Oat with NaOH) labelled with 58Fe given with 30 mL acai puree with honey

SUMMARY:
In the current study, the OAT fibril - Fe SA (Fe-oat 1) and OAT fibril - Fe NaOH (Fe-oat 2) will both be studied in vivo, alone are oat fibril powder add iron supplement is soluble in water and oat fibril powder add iron supplement is soluble in water in a food matrix (acai puree and honey) to assess their promise as Fe food fortificants.

This first in human study to bioavailability assessment and adverse effect of the OAT fibril - Fe SA (Fe-oat 1), OAT fibril - Fe NaOH (Fe-oat 2) and in a food matrix to assess their promise as Fe food fortificants.

This study will be conducted with the following objectives.

1. To conduct a stable Fe isotope study to evaluate the bioavailability of OAT-Fe formulated using two reducing agents (Fe-oat 1 and Fe-oat-2) and compared to FeSO4.
2. To compare the performance of Fe-oat 1 and 2 in a food matrix containing Fe inhibitors, (acai puree and honey) in comparison to FeSO4 in a similar meal matrix.

DETAILED DESCRIPTION:
Iron (Fe) deficiency is the most common nutrient deficiency present worldwide. Alternative solutions are needed for better absorption due to drawbacks that are associated with gastrointestinal side effects from Fe salt supplements. Additionally, Fe is difficult to add as a fortificant to foods due to the organoleptic changes that it causes. Reducing the particle size of iron salts improves their absorption, and submicron-sized Fe compounds are a promising solution in food matrices, although their tendency to oxidize and rapidly aggregate in solution limits their use in fortification.

A novel β-lactoglobulin (BLG) fibrils-Fe compound for use in Fe fortification was developed from milk proteins, and its evaluation in both in vitro digestion and in vivo (rat) bioavailability studies has been reported. It was observed that the material's reducing effect, colloidal stability, improved sensory performance and high bioavailability, making it promising for nutritional applications.

In the current study, a similar strategy is used to isolate amyloid fibrils from a vegan and more sustainable source, namely, oat protein. The reducing ability of the amyloid fibrils on the Fe salt - FeCl3 in the presence of sodium ascorbate (SA) or sodium hydroxide (NaOH), both food grade reagents, has shown the formation of a mixture of Fe2+ and Fe3+ particles with no observed aggregation. A previous human study showed that Fe3+ ions from submicron-sized ferric phosphate had a similar fractional Fe absorption (FIA) compared to that of ferrous sulfate (FeSO4), the current standard of care. The amyloid fibril systems by milk protein as efficient carriers for iron fortification. The evaluation in vitro digestion and in vivo bioavailability showed that β-lactoglobulin (β-lg) fibrils by milk protein disappeared 4 hours after providing this amyloid-rich supplement in the intestinal tract immediately. Moreover, the brain section of the mice supplemented with β-lg amyloid fibril showed no amyloid plague after 1 month of feeding. The β-lactoglobulin (β- lg) fibrils and plant-based oat share the same structure in the amyloid by milk protein. From these results, fibrils by oat are understood to be safe for nutrition.

Additionally, a recent study showed the possibility to produce amyloid fibrils from oat in full analogy to those obtained by BLG. In the current study, the OAT fibril - Fe SA (Fe-oat 1) and OAT fibril - Fe NaOH (Fe-oat 2) will both be studied in vivo, alone are oat fibril powder add iron supplement is soluble in water and oat fibril powder add iron supplement is soluble in water in a food matrix (acai puree and honey) to assess their promise as Fe food fortificants.

This first in human study to short-term food safety assessment and adverse effect of the OAT fibril - Fe SA (Fe-oat 1), OAT fibril - Fe NaOH (Fe-oat 2) and in a food matrix to assess their promise as Fe food fortificants.

The study will be a single-center, prospective cross-over study in which each subject receives 6 test conditions. The study will be conducted at the Institute of Nutrition, Mahidol University, Nakhon Pathom, Thailand. The study has been approved by the Ethical Board of Mahidol University and will be registered at www.clinicaltrials.gov. All subjects will provide written informed consent before any study procedures take place. During the screening, about 2 weeks before the start of the study, women will be assessed for eligibility. The study procedures will be explained to them in detail in a local language and following obtaining informed consent, a venipuncture blood sample (6 mL) will be collected for the determination of hemoglobin (Hb), serum ferritin (SF), c-reactive protein (CRP), thalassemia and pregnancy. Weight will be measured to the nearest 0.1 kg and height to the nearest 0.5 cm, to calculate BMI. An interview will be conducted to assess other inclusion and exclusion criteria. Women will be invited to screen until 52 eligible women have been enrolled to participate in the study. Each subject will complete the six iron absorption studies in which they will receive supplemental iron doses of 4 mg iron from the six products: (i) Fe-oat 1 alone, (ii) Fe-oat 1 with 30 mL acai puree with honey, (iii) Fe-oat 2 alone, (iv) Fe-oat 2 with 30 mL acai puree with honey, (v) FeSO4 alone, (vi) FeSO4 with 30 mL acai puree and honey. Polyphenol content of the acai puree will be measured at the Human Nutrition Laboratory.

The experimental phase will last for 37 days. The first three labeled iron doses will be administered on days 1, 3 and 5 between 07:00 and 09:00 in the morning after an overnight fast. After the third intervention, there will be a wait period of 14 days to allow for incorporation of the labeled iron into erythrocytes. On day 19, 21 and 23, the fourth, fifth and sixth intervention products will be given to the participants. It will be made sure that the randomization of the intervention products is done in such a manner that no two interventions with the same stable isotope are given to participants in the same week. Products 1, 3, and 5 from the list will be given in one week, and 2, 4 and 6 in the second week. There will be three blood sampling points excluding the screening: a baseline sampling on Day 1, sampling on day 17 and a final sampling 14 days after the fourth intervention product, on day 37, the last day of the study. These venous blood samples will be collected to determine Hb, SF and CRF, and erythrocyte isotopic enrichment.

Women will be randomized for the intervention administration order using a Python code. The participants will consume the labeled interventional products in the form of a solution under supervision of the investigators with or without the acai puree depending on the intervention type for the day. After consuming the test products, participants will refrain from eating or drinking for 3 h.

The Fe-oat 1 and Fe-oat 2 solutions will be produced at ETH Zurich at the Laboratory of Food and Soft Materials with food grade or pharmacopoeia grade chemicals and using 57Fe or 58Fe enriched elemental iron powders (Chemgas, Boulogne, France), and considering Good Manufacturing Practice regulations. The SOP for the preparation of the Fe-oat 1 and 2 will be provided upon request. The labelled FeSO4 solutions will be prepared at the Human Nutrition Laboratory (HNL) from 54Fe enriched elemental iron powders (Chemgas, Boulogne, France). The iron powders will be dissolved at room temperature in 1.7 M sulfuric acid (1.21 ml/100 mg Fe) in 100 ml HDPE bottles (Semadeni, Ostermundingen, Switzerland) flushed with argon. The resulting solutions will be brought to a concentration of 4 mg Fe/g solution with sterile pure water. The solutions will be divided into 1 g portions in PFA vials. The vials will be flushed with argon, tightly closed and kept at 4-8°C until use. The reagents will be of European Pharmacopoeia reagent grade (sulfuric acid 95-97%, Sigma-Aldrich, Buchs, Switzerland; Aqua ad iniect. B. Braun, Kantonsapotheke Zürich).

ELIGIBILITY:
Inclusion Criteria:

* female aged between 18-45 y old
* serum ferritin 10-50 μg/L
* hemoglobin ≥12g/dL
* BMI 18.5-24.9 kg/m2
* weight <70 kg
* signed informed consent
* able to communicate in and comprehend Thai language

Exclusion Criteria:

* anemia (Hb <12 g/dL)
* presence of thalassemia (with the exceptions of Hb E and alpha thal 1 trait)
* inflammation (CRP > 5 mg/L)
* chronic digestive, renal and/or metabolic disease
* chronic medications (except for oral contraceptives)
* use of vitamin, mineral and pre- and/or probiotic supplements in the previous 2 weeks before study initiation and during the course of the study
* blood transfusion, blood donation or significant blood loss over the past 4 months
* difficulties with blood sampling
* antibiotic treatment in the 4 weeks before study initiation
* pregnancy (tested in serum at screening) or intention to become pregnant
* lactation up to 6 weeks before study initiation
* earlier participation in a study using stable isotopes or participation in any clinical study within the last 30 days
* unable to comply with study protocol (e.g. not available on certain study appointment days or difficulties with blood withdrawal)
* inability to understand the information sheet and the informed consent form due to cognitive or language reasons
* smoking
* unwilling to use an effective method of contraception

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2023-04-03 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-02-29 (Actual)

PRIMARY OUTCOMES:
Fractional absorption of iron (%) | 37 days
  Fractional absorption of iron (%) from the iron supplements will be calculated based on the shift of the iron isotope ratios in the collected blood samples at least 14 days after the last administration of the isotopically labelled supplements.

SECONDARY OUTCOMES:
Hemoglobin (g/dL) | 37 days
  The determination of hemoglobin (g/dL) from blood sample
serum ferritin (ng/mL) | 37 days
  The determination of serum ferritin (ng/mL) from blood sample
c-reactive protein (mg/L) | 37 days
  The determination of c-reactive protein (mg/L) from blood sample

CONTACTS AND LOCATIONS:
Overall Officials: Sueppong Gowachirapant, Principal Investigator — Mahidol University
Locations (1):
- Institute of Nutrition, Institute of Nutrition Mahidol University, Salaya, Changwat Nakhon Pathom, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Miller JL. Iron deficiency anemia: a common and curable disease. Cold Spring Harb Perspect Med. 2013 Jul 1;3(7):a011866. doi: 10.1101/cshperspect.a011866. PMID 23613366
- [Background] Tolkien Z, Stecher L, Mander AP, Pereira DI, Powell JJ. Ferrous sulfate supplementation causes significant gastrointestinal side-effects in adults: a systematic review and meta-analysis. PLoS One. 2015 Feb 20;10(2):e0117383. doi: 10.1371/journal.pone.0117383. eCollection 2015. PMID 25700159
- [Background] Allen L, De Benoist B, Dary O, Hurrell R. Guidelines on food fortification with micronutrients: JSTOR; 2006.
- [Background] Hurrell RF. Fortification: overcoming technical and practical barriers. J Nutr. 2002 Apr;132(4 Suppl):806S-12S. doi: 10.1093/jn/132.4.806S. PMID 11925486
- [Background] Acosta E. Bioavailability of nanoparticles in nutrient and nutraceutical delivery. Current opinion in colloid & interface science. 2009;14(1):3-15.
- [Background] Hilty FM, Arnold M, Hilbe M, Teleki A, Knijnenburg JT, Ehrensperger F, Hurrell RF, Pratsinis SE, Langhans W, Zimmermann MB. Iron from nanocompounds containing iron and zinc is highly bioavailable in rats without tissue accumulation. Nat Nanotechnol. 2010 May;5(5):374-80. doi: 10.1038/nnano.2010.79. Epub 2010 Apr 25. PMID 20418865
- [Background] Rohner F, Ernst FO, Arnold M, Hilbe M, Biebinger R, Ehrensperger F, Pratsinis SE, Langhans W, Hurrell RF, Zimmermann MB. Synthesis, characterization, and bioavailability in rats of ferric phosphate nanoparticles. J Nutr. 2007 Mar;137(3):614-9. doi: 10.1093/jn/137.3.614. PMID 17311949
- [Background] Huber DL. Synthesis, properties, and applications of iron nanoparticles. Small. 2005 May;1(5):482-501. doi: 10.1002/smll.200500006. PMID 17193474
- [Background] Shen Y, Posavec L, Bolisetty S, Hilty FM, Nystrom G, Kohlbrecher J, Hilbe M, Rossi A, Baumgartner J, Zimmermann MB, Mezzenga R. Amyloid fibril systems reduce, stabilize and deliver bioavailable nanosized iron. Nat Nanotechnol. 2017 Jul;12(7):642-647. doi: 10.1038/nnano.2017.58. Epub 2017 Apr 24. PMID 28436960
- [Background] Baumgartner J, Winkler HC, Zandberg L, Tuntipopipat S, Mankong P, Bester C, Hilty F, Zeevaart JR, Gowachirapant S, Zimmermann MB. Iron from nanostructured ferric phosphate: absorption and biodistribution in mice and bioavailability in iron deficient anemic women. Sci Rep. 2022 Feb 18;12(1):2792. doi: 10.1038/s41598-022-06701-x. PMID 35181698
- [Background] Zhou J, Li T, Peydayesh M, Usuelli M, Lutz-Bueno V, Teng J, Wang L, Mezzenga R. Oat Plant Amyloids for Sustainable Functional Materials. Adv Sci (Weinh). 2022 Feb;9(4):e2104445. doi: 10.1002/advs.202104445. Epub 2021 Dec 20. PMID 34931493
- [Background] Cercamondi CI, Egli IM, Mitchikpe E, Tossou F, Zeder C, Hounhouigan JD, Hurrell RF. Total iron absorption by young women from iron-biofortified pearl millet composite meals is double that from regular millet meals but less than that from post-harvest iron-fortified millet meals. J Nutr. 2013 Sep;143(9):1376-82. doi: 10.3945/jn.113.176826. Epub 2013 Jul 24. PMID 23884388
- [Background] BROWN E, HOPPER J Jr, HODGES JL Jr, BRADLEY B, WENNESLAND R, YAMAUCHI H. Red cell, plasma, and blood volume in the healthy women measured by radiochromium cell-labeling and hematocrit. J Clin Invest. 1962 Dec;41(12):2182-90. doi: 10.1172/JCI104677. No abstract available. PMID 14015940
- [Background] International Nutritional Anemia Consultative Group (INACG) WHOW, United Nations Childrens Fund (UNICEF). Guidelines for the use of iron supplements to prevent and treat iron deficiency anemia. 1998.
- [Background] von Moos LM, Schneider M, Hilty FM, Hilbe M, Arnold M, Ziegler N, Mato DS, Winkler H, Tarik M, Ludwig C, Naegeli H, Langhans W, Zimmermann MB, Sturla SJ, Trantakis IA. Iron phosphate nanoparticles for food fortification: Biological effects in rats and human cell lines. Nanotoxicology. 2017 May;11(4):496-506. doi: 10.1080/17435390.2017.1314035. Epub 2017 Apr 20. PMID 28368214